CLINICAL TRIAL: NCT06478407
Title: Community Screening Study of Diabetic Retinopathy in Tianjin in 2024
Acronym: CSSODRIT
Status: Recruiting | Type: Observational
Sponsor: Li Xiaorong (Other)
Collaborators: Tianjin Medical University Eye Hospital (Other)
Responsible Party: Sponsor-Investigator, Li Xiaorong, PROFESSOR, Tianjin Medical University Eye Hospital
Organization: Tianjin Medical University Eye Hospital (Other)
Other Study IDs: 2024
Record Dates: First submitted 2024-06-22; First posted 2024-06-27 (Actual); Last update posted 2024-07-10 (Actual); Status verified 2024-07

CONDITIONS: Diabetic Retinopathy
Keywords: diabetic retinopathy
MeSH Terms: conditions — Diabetic Retinopathy

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples With DNA — Blood and Midstream clean urine
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Diabetic retinopathy screening group: Diabetes patients in the community to accept unified eye test, confirm whether patients with diabetic retinopathy

SUMMARY:
Through this study, the investigators hope to understand the prevalence and influencing factors of diabetic retinopathy in Tianjin, improve the ability of complication detection and intervention in diabetic patients in primary medical and health institutions, and build a diabetes prevention and treatment network. The investigators should adhere to the policy of prevention first, combined with prevention and control, and explore a diabetes' prevention and control model suitable for our city. Extensive publicity and education should be carried out to improve the awareness of self-management ，improve the screening rate of diabetic retinopathy, and reduce the blindness rate.

DETAILED DESCRIPTION:
West of the city, and hebei, heping and binhai new area to carry out the work, diabetic retinopathy screening on 18000 diabetic patients in fundus examination. Tianjin medical university eye hospital, project team, formed in grassroots medical institutions are responsible for screening fundus examination in patients with diabetes, related inspection including vision, computer optometry, fundus photography and optical coherence tomography angiography (OCTA), etc. Blood samples were collected from patients in Hexi District and Heping District to detect glycosylated hemoglobin. Glycated albumin, urine ACR and CO breath test were performed in Chu Hsien-I Memorial Hospital of Tianjin Medical University. Health records were established for the screening personnel after the examination

ELIGIBILITY:
Inclusion Criteria:

- 1: Clear awareness, barrier-free communication

2: diabetes

Exclusion Criteria:

* 1: Have left the registered home address

  2: In the last 6 months, you have not lived in your place of residence

  3: Have a serious mental illness

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients with diabetes receive a unified eye examination in the community to confirm whether they have diabetic retinopathy
Sampling Method: Non-Probability Sample
Enrollment: 18000 (Estimated)
Dates: Start 2024-03-28 (Actual); Primary Completion 2025-03-28 (Estimated); Study Completion 2025-03-28 (Estimated)

PRIMARY OUTCOMES:
Classification of diabetic retinopathy | At screening
  Fundus images were taken by fundus camera and graded

SECONDARY OUTCOMES:
blood routine examination | At screening
  Blood was collected and tested
OCTA imaging indicators | At screening
  OCTA machine was used to photograph the fundus
blood biochemistry | At screening
  Blood was collected and tested
glycosylated hemoglobin | At screening
  Blood was collected and tested
glycated albumin | At screening
  Blood was collected and tested
Urine ACR | At screening
  Urine was collected and tested
Blood vessel color Doppler ultrasound of extremities | At screening
  Blood vessels of extremities were photographed by color Doppler ultrasound

CONTACTS AND LOCATIONS:
Overall Officials: Xiaorong Li, professor, Principal Investigator — Tianjin Medical University Eye Hospital
Locations (1):
- Tianjin Medical University Eye Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol (2024-01-26): https://cdn.clinicaltrials.gov/large-docs/07/NCT06478407/Prot_000.pdf
  • Informed Consent Form (2024-01-29): https://cdn.clinicaltrials.gov/large-docs/07/NCT06478407/ICF_001.pdf